CLINICAL TRIAL: NCT03888924
Title: Bacille Calmette-Guérin (BCG) Vaccine In Radiologically Isolated Syndrome (RIS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Ristori, Medical director, PhD, S. Andrea Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCG-RIS-01
Record Dates: First submitted 2018-09-04; First posted 2019-03-25 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: BCG Vaccine; Radiologically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: This is a phase II, double blind, randomized, controlled, multicenter study with two parallel groups of subjects.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In order to guarantee a double blind design, participants, assessing neurologists and neuroradiologists will be masked to treatment allocation. A "two-physician-treating and assessing-model" will be used
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG treated patients (Experimental): a single dose of Bacille Calmette-Guerin vaccine
  Interventions: Drug: Bacille Calmette-Guerin vaccine
- Placebo treated patients (Placebo Comparator): a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bacille Calmette-Guerin vaccine — One dose (0.1 mL) contains 50 μg of the semi-dry mass of BCG bacilli, i.e. from 150,000 to 600,000 of live BCG bacilli (Bacillus Calmette-Guerin), the Brazilian Moreau substrain.
  One ampoule or vial with the powder contains: 0.5 mg (from 1.5 mln to 6 mln) of live BCG bacilli (Bacillus Calmette-Guerin), the Brazilian Moreau substrain.
  Powder: monosodium glutamate. Solvent: isotonic solution of sodium chloride.
  Other Names: BCG 10 Anti-Tuberculosis Vaccine
  Arms: BCG treated patients
Drug: Placebo — isotonic solution of sodium chloride (2mL vials).
  Arms: Placebo treated patients

SUMMARY:
Multiple sclerosis (MS) witnessed relevant therapeutic progress in the last decade. Following the extraordinary progress in the treatment of relapsing-remitting (RR) multiple sclerosis (MS), two major unmet needs remain to be addressed by translational research in this field: progressive MS and the "dream" of a world free of MS. As far as the latter is concerned, the investigators can hope to make the dream come true by understanding the etiology of the disease and hence design definitive cures. A more realistic and pragmatic perspective may be the prevention of the clinical onset of the disease, a research field that promises to become increasingly important as the integration of genetic data with endophenotypes, magnetic resonance imaging and other biomarkers ameliorates the ability to predict the development of the disease under clinical circumstance. Bacille Calmette-Guerin (BCG) vaccine has been tested with encouraging results in early MS and clinically isolated syndrome (CIS). The knowledge that disease-modifying therapies work best when used early in the demyelinating process raises the question about whether to try this approach - which is safe, cheap and handy - in individuals with radiologically isolated syndrome (RIS).

Radiologically isolated syndrome is a new entity, diagnosed when the unanticipated magnetic resonance imaging (MRI) finding of brain spatial dissemination of focal white matter (WM) lesions highly suggestive of MS occurs in subjects without symptoms of MS, and with normal neurological examinations. Conversion to clinically isolated syndromes (CIS) were described in 84% of RIS individuals with spinal cord lesions over a median time of 1.6 years from the date of the first MRI. Whether or not to treat this condition remains currently a clinical conundrum. Bacille Calmette-Guérin (BCG) vaccine may have these characteristics since it resulted beneficial in early MS and first demyelinating episodes. Being safe, cheap and handy, the investigators propose to investigate its use to prevent progression of the demyelinating process in radiologically isolated syndrome. An approach such as BCG vaccine seems appropriate as a front-line immunomodulatory approach for RIS people. In a pilot study BCG vaccine was safe and effective in reducing disease activity at MRI, and the risk of developing persistent T1-hypointense lesions ('black holes' -BH- expression of tissue damage) in subjects with MS.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) witnessed relevant therapeutic progress in the last decade. This notwithstanding, safety, quality of life and overtreatment remain elements of strong concern for the subjects. Safe and manageable therapies that can be used since the (biological) onset of the disease, without risk of overtreatment, are important unmet needs in MS.

Following the extraordinary progress in the treatment of relapsing-remitting (RR) multiple sclerosis (MS), two major unmet needs remain to be addressed by translational research in this field: progressive MS and the "dream" of a world free of MS. As far as the latter is concerned, the investigators can hope to make the dream come true by understanding the etiology of the disease and hence design definitive cures. Unfortunately this perspective is neither at hand, nor it can be taken for granted that the etiologic targets, once discovered, will be readily treatable.

A more realistic and pragmatic perspective may be the prevention of the clinical onset of the disease, a research field that promises to become increasingly important as the integration of genetic data with endophenotypes, magnetic resonance imaging and other biomarkers ameliorates the ability to predict the development of the disease under clinical circumstance.

Epidemiological data supporting vitamin D supplementation and smoking avoidance are candidate approaches for primary and secondary prevention of the disease. Among other interventions that may have characteristics compatible with those of a preventive treatment, Bacille Calmette-Guerin (BCG) vaccine has been tested with encouraging results in early MS and clinically isolated syndrome (CIS). The knowledge that disease-modifying therapies work best when used early in the demyelinating process raises the question about whether to try this approach - which is safe, cheap and handy - in individuals with radiologically isolated syndrome (RIS).

Radiologically isolated syndrome is a new entity, diagnosed when the unanticipated magnetic resonance imaging (MRI) finding of brain spatial dissemination of focal white matter (WM) lesions highly suggestive of MS occurs in subjects without symptoms of MS, and with normal neurological examinations. Approximately one-third and two-thirds of individuals experience respectively clinical onset and/or radiological progression over a mean follow-up of five years. However, predictors (male sex, age < 37, spinal cord involvement) of higher risk of progression have been identified and conversion to clinically isolated syndromes (CIS) were described in 84% of RIS individuals with spinal cord lesions over a median time of 1.6 years from the date of the first MRI; the same predictors have recently been shown to precede evolution toward primary progressive MS. Whether or not to treat this condition remains currently a clinical conundrum.

Bacille Calmette-Guérin (BCG) vaccine may have these characteristics since it resulted beneficial in early MS and first demyelinating episodes. Being safe, cheap and handy, the investigators propose to explore its use to prevent progression of the demyelinating process in radiologically isolated syndrome.

An approach such as BCG vaccine seems appropriate as a front-line immunomodulatory approach for RIS people. This project is proposed in the context of the activity of the Center for Experimental Neurological Therapies (CENTERS - a special project by the Fondazione Italiana Sclerosi Multipla - FISM). CENTERS is especially dedicated to phase II trials of this nature (independent, repurposing studies, that may be only funded by not-for-profit institutions).

1.2 Preliminary Results

Experimental and epidemiological evidences suggested benefit of exposure to microbial products (in the absence of infection, as is the case of vaccinations) in autoimmunity, including MS. In a pilot study BCG vaccine was safe and effective in reducing disease activity at MRI, and the risk of developing persistent T1-hypointense lesions ('black holes' -BH- expression of tissue damage) in subjects with MS. A placebo-controlled trial in people with clinically isolated syndrome supported the findings of the pilot study. The researchers observed benefit on disease activity at MRI, reduced development of BH, benefit on conversion to clinically definite MS over 5 years, during which the subjects took interferon beta beginning from six months after BCG or placebo.

The investigators consider timely an extension of the adjuvant approach to subjects with RIS, also considering recent achievements in 'metrics' suitable to analyze this condition: neuroimaging has recently allowed to improve the characterization of RIS (including the identification of individuals at higher risk of progression to MS; and to disclose cortical lesions and axonal damage in RIS brain; immune-metabolic profiling provides a complex correlation between immunometabolic cellular variables, that seems especially apt to analyze preclinical phase of neuroinflammation and to study an approach whose underlying mechanisms of actions remain largely unknown, in spite of encouraging clinical results.

1.3 Scientific rationale and main objectives

BCG vaccine showed beneficial effects on disease activity and possibly on tissue damage in relapsing-remitting MS and clinically isolated syndrome. The investigators now propose to evaluate whether and how BCG vaccine exerts favorable biological effects in individuals with RIS.

At present it is unclear whether the neuroprotective/neurorepair potential of BCG is a consequence of its ability to reduce central nervous system (CNS) inflammation or it depends on additional and specific mechanisms. Notably, neuroprotection after BCG vaccination was reported in models of Parkinson disease, suggesting a neuroprotective vaccine paradigm in which general (nonself-reactive) immune stimulation in the periphery can limit potentially deleterious microglial responses to a neuronal insult. Accordingly, convergent evidences suggest a role of BCG, as tumor necrosis factor (TNF)-inducer, in another immune-mediated disease, type I diabetes: TNF receptor 2 may mediate, at least in part, beneficial effects of BCG in neuroinflammation and type 1 diabetes by favoring apoptosis of autoreactive T cells, counteracting T cell regulatory deficit and last, but not least, fostering tissue repair.

Metabolic abnormalities suggestive of axonal damage were reported in a substantial proportion of RIS subjects and cortical lesions of fronto-temporal lobes were associated with predictors of evolution to multiple sclerosis (MS), such as spinal cord involvement, presence of oligoclonal bands on cerebrospinal fluid and dissemination in time on brain MRI. The researchers aim at verifying potential beneficial effects of BCG vaccination in people with RIS, evaluating MRI metrics of macroscopic brain damage, as well as subtle tissue damage as assessed by both conventional and non conventional MRI techniques. On the immunological side the investigators will assess the immune-metabolic status of RIS people as well as their regulatory T cell potential: a multiple parameter analysis will provide a meta-immunologic profiling that has been recently shown to be impaired in MS. This will be aimed at creating a follow-up scheme which should allow to monitor RIS people over time, before and after BCG vaccine.

To reach the above purposes the investigators propose a 3 years longitudinal study project, considered appropriate taking into account the relative rarity of RIS condition as well as the need of an adequate follow-up to obtain informative outcome measures (see methods).

The groups that engendered the above achievements are collaborators of this project, thus warranting the experience and competence to pursue the proposed research.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female of any race and > 18 years old.
2. Diagnosis of RIS (4) within the last five years.
3. Signed Informed Consent.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Concomitant or previous use of immunosuppressive or immunomodulating treatment (except sporadic use of corticosteroids) within the last five years.
3. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation. Such conditions may include cardiovascular, pulmonary, hepatic, renal, severe systemic mycotic infections, metabolic diseases or malignancies, primary or secondary immunodeficiencies as determined by medical history, physical exam, laboratory tests, chest X-ray, electrocardiogram (ECG), and Mantoux reaction.
4. Any medical or psychiatric condition that may affect the subjects ability to give informed consent, or to complete the study, or if the subject is considered by the treating neurologist to be, for any other reason, an unsuitable candidate for this study.
5. Subjects with inability to successfully undergo MRI scans.
6. Concomitant radiotherapy.
7. Known hypersensitivity to any component of the vaccine.
8. Past bone marrow stem cell transplantation and organ transplantation.
9. Other vaccinations in the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
cumulative number of CUAL (new gadolinium T1-weighted lesions and non-enhancing new and newly enlarging T2-weighted lesions) on MRI scans over 1 year. | 12 months
  To evaluate the cumulative number of new combined unique active lesions (CUAL; defined as new gadolinium T1-weighted lesions and non-enhancing new and newly enlarging T2-weighted lesions) on magnetic resonance imaging (MRI) scans over 1 year.
  Brain MRI will be acquired in all subjects at each centre using a magnet at 1.5T or 3T.
  * A sagittal survey image will be used to identify the anterior and posterior commissure (AC and PC).
  * A dual-echo, turbo spin-echo sequence (slice thickness: 3mm).
  * A high-resolution (3D, MPRAGE) T1- weighted image (slice thickness: 1mm).
  * A Magnetization Transfer (MT) sequence will be performed acquiring two 2-dimensional gradient-echo sequences, one without and one with MT saturation pulse (slice thickness: 3 mm).
  * A double inversion recovery (DIR) sequence
  * A T1-weighted scan, post-gadolinium injection, after 10-minute wait period.
  * A FLAIR sequence to be acquired between the DIR and the T1-weighted scans, after the gadolinium injection.

SECONDARY OUTCOMES:
Time to the first clinical event. | 36 months
  The secondary endpoint will be the time to the first clinical event over the 3 years period.
  Five visits (including physical and neurological examinations) per subject are planned:
  * Visit 1 - from day -3 to day +1
  * Visit 2 - 6 months (±7 days)
  * Visit 3 - 12 months (±7 days)
  * Visit 4 - 24 months (±7 days)
  * Visit 5 - 36 months (±7 days)

OTHER OUTCOMES:
number of cortical lesions | 6, 12, 24, 36 months
  To evaluate the number of cortical lesions on magnetic resonance imaging (MRI) scans at 6 months, as well as at 1, 2 and 3 years: Cortical lesions will be assessed on the DIR sequence and defined as those focal hyperintensities entirely or partly located in the cortical GM.
Percentage of Brain Volume Changes (PBVC) | 6, 12, 24, 36 months
  Brain atrophy (global and regional) will be assessed on the 3D T1-weighted images using the software SIENA/SIENAX (Structural Image Evaluation, using Normalization, of Atrophy) method.
Cortical and white matter Volume Changes | 6, 12, 24, 36 months
  Brain atrophy (global and regional) will be assessed on the 3D T1-weighted images using the software SIENA/SIENAX (Structural Image Evaluation, using Normalization, of Atrophy) method. To avoid GM misclassification due to WM lesions, the latter will be masked out and refilled with intensities matching the surrounding normal-appearing WM before segmentation analysis. Volume in the subcortical grey matter will be assessed with FMRIB's Integrated Registration and Segmentation Tool (FIRST).
Magnetization Transfer ratio (MTr) in lesions | 6, 12, 24, 36 months
  Magnetization Transfer (MT) sequence will be performed acquiring two 2-dimensional gradient-echo sequences, one without and one with MT saturation pulse, which allows to obtain MT ratio in lesions, and normal-appearing brain.
Magnetization Transfer ratio (MTr) in normal-appearing brain | 6, 12, 24, 36 months
  Magnetization Transfer (MT) sequence will be performed acquiring two 2-dimensional gradient-echo sequences, one without and one with MT saturation pulse, which allows to obtain MT ratio in lesions, and normal-appearing brain.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ristori, Principal Investigator — S.Andrea Hospital, University of Roma La Sapienza
Locations (1):
- Center for Experimental Neurological Therapies (CENTERS), S. Andrea Hospital, Faculty of Medicine and Psychology, "Sapienza" University of Rome, Rome, Italy